CLINICAL TRIAL: NCT07284927
Title: Clinical Study of LV009 Injection for the Treatment of Relapsed/Refractory CD19-Positive Hematologic and Lymphoid Malignancies
Brief Title: Clinical Study of LV009 Injection for the Treatment of Hematologic and Lymphoid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-012-3
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LV009 Injection (Experimental)
  Interventions: Biological: LV009 Injection

INTERVENTIONS:
Biological: LV009 Injection — Eligible subjects who pass the screening process after providing signed informed consent will receive an infusion of LV009 Injection.

SUMMARY:
This clinical trial is designed as a single-arm, open-label, single-center, investigator-initiated, early-phase study. Its primary objective is to evaluate the safety of LV009 Injection in subjects with relapsed/refractory CD19-positive hematolymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years (inclusive), irrespective of sex and race.
2. Life expectancy greater than 12 weeks.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 2.
4. Meets the National Comprehensive Cancer Network (NCCN) criteria for relapsed or refractory disease, with a confirmed diagnosis of CD19-positive hematolymphoid malignancy
5. Adequate hepatic, renal, and cardiopulmonary function
6. Absolute lymphocyte count (ALC) ≥ 0.5 × 10⁹/L; Platelet count ≥ 50 × 10⁹/L; CD3-positive T-cell count ≥ 150 cells/μL

Exclusion Criteria:

1. Patients who, in the investigator's judgment at screening, require long-term use of immunosuppressive agents.
2. History of cerebrovascular accident or convulsive seizures within 6 months prior to signing the informed consent form.
3. Presence of other active malignant diseases besides the disease under study, with the exception of carcinoma in situ.
4. Patients with severe cardiac disease, unstable systemic diseases, or chronic progressive neurological disorders, etc.
5. Patients who have received CAR-T therapy or other genetically modified cell therapies prior to screening.
6. Patients who have participated in other clinical studies within 1 month prior to screening.
7. Evidence of central nervous system involvement at the time of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Safety | 2 years
  Adverse Events Occurring During the Treatment Period (TEAEs), Serious Adverse Events (SAEs), Replication-Competent Lentivirus (RCL), and Lentiviral Insertion Site Status (Assessed according to the Common Terminology Criteria for Adverse Events, Version 5.0, NCI CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No